CLINICAL TRIAL: NCT02396901
Title: Goal Direct Therapy to Prevent Acute Kidney Injury After Cardiac Surgery
Brief Title: Goal Direct Therapy to Prevent Acute Kidney Injury
Acronym: GDT-AKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduesley Santana Santos, RN, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDC 4163/14/143
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Acute Kidney Injury
Keywords: early goal direct therapy; preventive strategies; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GDT group (Experimental): Patients randomized to the GDT Group will care from a protective strategy with the suspension of angiotensin-converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARB) 48 hours before surgery and receive hydration with lactated Ringer's solution at the rate of 1 mL/kg/h in the night before the surgery until the surgical procedure and perioperative hemodynamic therapy.
  Interventions: Other: Goal Direct Therapy
- Control group (Placebo Comparator): Patients randomized to the control group will be treated in accordance with the care in the institution's routine.

INTERVENTIONS:
Other: Goal Direct Therapy — Goal Direct Therapy - in this group patients will receive the standard treatment according with institutional protocol.
  Arms: GDT group

SUMMARY:
This is an randomised controlled trial to investigate an strategy based in a protocol in prevention of acute kidney injury after cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial to assess the influence of use of angiotensin-converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARB) in the development of the Acute Kidney Injury in the postoperative period of cardiac surgery. Patients undergoing cardiac surgery at the Heart Institute (InCor) - Brazil, will be randomized and in accordance with a list of random numbers, generated by a computer program, will be allocated in one of the groups (GDT or standard).

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with Cardiopulmonary Bypass (CPB); Age greater than 18 years; Chronic kidney disease stages 3 and 4 (GFR less than 60 mL/min and greater than 15 mL/min); Sign the informed consent form.

Exclusion Criteria:

* Chronic renal insufficiency (GFR less than 15 mL/min); Heart surgery without CPB; Aortic procedures; Heart transplant or congenital heart disease; Prior use of Intra-Aortic Balloon Pump; Decompensated heart failure; Participation in other research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 48h after cardiac surgery
  Development of acute kidney injury according to AKIN (Acute Kidney Injury Network) criterion.

SECONDARY OUTCOMES:
Serious clinical complications | For 28 days
  Defined according to the guidelines of the Society of Thoracic Surgeons and include: stroke, need for invasive mechanical ventilation for more than 48 hours, mediastinitis, or deep infection of the surgical wound, mortality, need for reoperation.

REFERENCES:
- [Background] Liano F, Pascual J. Epidemiology of acute renal failure: a prospective, multicenter, community-based study. Madrid Acute Renal Failure Study Group. Kidney Int. 1996 Sep;50(3):811-8. doi: 10.1038/ki.1996.380. PMID 8872955
- [Background] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1--coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S2-22. doi: 10.1016/j.athoracsur.2009.05.053. PMID 19559822
- [Result] Mangano CM, Diamondstone LS, Ramsay JG, Aggarwal A, Herskowitz A, Mangano DT. Renal dysfunction after myocardial revascularization: risk factors, adverse outcomes, and hospital resource utilization. The Multicenter Study of Perioperative Ischemia Research Group. Ann Intern Med. 1998 Feb 1;128(3):194-203. doi: 10.7326/0003-4819-128-3-199802010-00005. PMID 9454527
- [Result] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670
- [Result] Conlon PJ, Stafford-Smith M, White WD, Newman MF, King S, Winn MP, Landolfo K. Acute renal failure following cardiac surgery. Nephrol Dial Transplant. 1999 May;14(5):1158-62. doi: 10.1093/ndt/14.5.1158. PMID 10344355
- [Result] Bahar I, Akgul A, Ozatik MA, Vural KM, Demirbag AE, Boran M, Tasdemir O. Acute renal failure following open heart surgery: risk factors and prognosis. Perfusion. 2005 Oct;20(6):317-22. doi: 10.1191/0267659105pf829oa. PMID 16363316
- [Result] Boldt J, Brenner T, Lang J, Kumle B, Isgro F. Kidney-specific proteins in elderly patients undergoing cardiac surgery with cardiopulmonary bypass. Anesth Analg. 2003 Dec;97(6):1582-1589. doi: 10.1213/01.ANE.0000090146.02929.2E. PMID 14633524 (Retraction: PMID 21451070 Anesth Analg. 2011 May;112(5):1146)
- [Result] Fleming I, Hecker M, Busse R. Intracellular alkalinization induced by bradykinin sustains activation of the constitutive nitric oxide synthase in endothelial cells. Circ Res. 1994 Jun;74(6):1220-6. doi: 10.1161/01.res.74.6.1220. PMID 7514511
- [Result] Burns KE, Chu MW, Novick RJ, Fox SA, Gallo K, Martin CM, Stitt LW, Heidenheim AP, Myers ML, Moist L. Perioperative N-acetylcysteine to prevent renal dysfunction in high-risk patients undergoing cabg surgery: a randomized controlled trial. JAMA. 2005 Jul 20;294(3):342-50. doi: 10.1001/jama.294.3.342. PMID 16030279
- [Result] Fisher AR, Jones P, Barlow P, Kennington S, Saville S, Farrimond J, Yacoub M. The influence of mannitol on renal function during and after open-heart surgery. Perfusion. 1998 May;13(3):181-6. doi: 10.1177/026765919801300305. PMID 9638715
- [Result] Hynninen MS, Niemi TT, Poyhia R, Raininko EI, Salmenpera MT, Lepantalo MJ, Railo MJ, Tallgren MK. N-acetylcysteine for the prevention of kidney injury in abdominal aortic surgery: a randomized, double-blind, placebo-controlled trial. Anesth Analg. 2006 Jun;102(6):1638-45. doi: 10.1213/01.ANE.0000219590.79796.66. PMID 16717300
- [Result] Benedetto U, Sciarretta S, Roscitano A, Fiorani B, Refice S, Angeloni E, Sinatra R. Preoperative Angiotensin-converting enzyme inhibitors and acute kidney injury after coronary artery bypass grafting. Ann Thorac Surg. 2008 Oct;86(4):1160-5. doi: 10.1016/j.athoracsur.2008.06.018. PMID 18805152
- [Result] Rosner MH, Okusa MD. Acute kidney injury associated with cardiac surgery. Clin J Am Soc Nephrol. 2006 Jan;1(1):19-32. doi: 10.2215/CJN.00240605. Epub 2005 Oct 19. PMID 17699187
- [Result] Bakris GL, Weir MR. Angiotensin-converting enzyme inhibitor-associated elevations in serum creatinine: is this a cause for concern? Arch Intern Med. 2000 Mar 13;160(5):685-93. doi: 10.1001/archinte.160.5.685. PMID 10724055
- [Result] Thakar CV, Arrigain S, Worley S, Yared JP, Paganini EP. A clinical score to predict acute renal failure after cardiac surgery. J Am Soc Nephrol. 2005 Jan;16(1):162-8. doi: 10.1681/ASN.2004040331. Epub 2004 Nov 24. PMID 15563569
- [Result] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 3--valve plus coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S43-62. doi: 10.1016/j.athoracsur.2009.05.055. PMID 19559824